CLINICAL TRIAL: NCT05083793
Title: The Effect of Pregabalin on Post-operative Pain and Opioid Consumption in Spine Surgery, a Prospective, Randomized, Controlled Study
Brief Title: the Effect of Pregabalin on Postoperative Pain and Opioid Consumption in Spine Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Professor of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17101526
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
Keywords: pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: care provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): patients have spine surgery receive oral pregabalin 150 mg 1 hour before surgery
  Interventions: Drug: Pregabalin 150mg
- Placebo group (Placebo Comparator): patients will receive placebo 1 hour before surgery with a sip of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin 150mg — The effect of pregabalin on post-operative pain
  Other Names: Pregabalin
  Arms: Study group
Other: Placebo — patients will receive placebo one hour before operation
  Arms: Placebo group

SUMMARY:
The effect of pregabalin on post-operative pain and opioid consumption in spine surgery, a prospective, randomized, controlled study

DETAILED DESCRIPTION:
Aim of the work:

The aim of our study is to compare the analgesic effect of pre-emptive oral pregabalin 150mg on acute postoperative pain and opioid consumption in spine surgery. Evaluated by visual analog scale (VAS)

primary outcome measure is the total amount of rescue morphine received by patients for 24h postoperatively.

secondary outcome measures include level of acute postoperative pain by VAS, and duration of hospital stay

Patients and methods :

This study will be carried out after being approved from the Medical Research Ethical Committee, Faculty of Medicine, Assiut University, Assiut, Egypt, and after obtaining a written informed consents from all participating patients.

inclusion criteria: This prospective randomized clinical study will include eighty patients with ASA I-II, aged 18-60 years scheduled for spine surgery

Exclusion criteria : Excluded from the study are patients with known allergy to the study drugs, significant cardiac, respiratory, renal, CNS or hepatic disease, drug or alcohol abuse, pregnant women, patients refusing participation and psychiatric or mental illness that would interfere with perception and assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* : This prospective randomized clinical study will include eighty patients with ASA I-II, aged 18-60 years scheduled for spine surgery

Exclusion Criteria:

* : Excluded from the study are patients with known allergy to the study drugs, significant cardiac, respiratory, renal, CNS or hepatic disease, drug or alcohol abuse, pregnant women, patients refusing participation and psychiatric or mental illness that would interfere with perception and assessment of pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Morphia dose | 24 hour postoperative
  the total amount of rescue morphine received by patients for 24h postoperatively.

SECONDARY OUTCOMES:
Postoperative pain | 24 hour postoperative
  post operative VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Maher, MD, Study Chair — Assiut University Hospitals
Locations (1):
- Mahmoud Maher, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
make individual participant data (IPD) available to other researchers
Supporting Information: Study Protocol
Time Frame: one year
Access Criteria: Study protocol
URL: https://pubmed.ncbi.nlm.nih.gov/15315511/

REFERENCES:
- [Background] Ben-Menachem E. Pregabalin pharmacology and its relevance to clinical practice. Epilepsia. 2004;45 Suppl 6:13-8. doi: 10.1111/j.0013-9580.2004.455003.x. PMID 15315511
- [Background] Hindmarch I, Trick L, Ridout F. A double-blind, placebo- and positive-internal-controlled (alprazolam) investigation of the cognitive and psychomotor profile of pregabalin in healthy volunteers. Psychopharmacology (Berl). 2005 Dec;183(2):133-43. doi: 10.1007/s00213-005-0172-7. Epub 2005 Nov 9. PMID 16205916
- [Background] Sebastian B, Talikoti AT, Nelamangala K, Krishnamurthy D. Effect of Oral Pregabalin as Preemptive Analgesic in Patients Undergoing Lower Limb Orthopedic Surgeries under Spinal Anaesthesia. J Clin Diagn Res. 2016 Jul;10(7):UC01-4. doi: 10.7860/JCDR/2016/18854.8081. Epub 2016 Jul 1. PMID 27630927
- See also: Pregabalin pharmacology and its relevance to clinical practice — https://pubmed.ncbi.nlm.nih.gov/15315511/